CLINICAL TRIAL: NCT06576895
Title: Nutrition Practice in Critically Ill Adults - an Observational Study
Brief Title: Nutrition Practice in Critically Ill Adults
Acronym: NUTRIENT
Status: Recruiting | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: ANZIC-RC/ER002
Record Dates: First submitted 2024-08-14; First posted 2024-08-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-08

CONDITIONS: Critical Illness
Keywords: Intensive Care; Nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To determine the role of nutrition in recovery from critical illness, current practice must first be understood. However, no benchmarking process currently exists for nutrition practice during critical illness, from ICU admission to hospital discharge. This vital gap requires addressing.

The aim of this study is to inform and re-design models of nutrition care and generate research priorities for the future by obtaining data on nutrition provision and practice and that of consumer preference for nutrition care.

DETAILED DESCRIPTION:
This study is a multi-centre observational study of nutrition practices in critically ill adults across ANZ. Two study periods are proposed, the first confirmed period in Q3-2024 and the second in 2026.

This study is part of a larger study which consists of three interconnected streams. This study forms part of Stream 2 which is about understanding nutrition practice and provision in adults with critical illness. The findings from this study will be used to inform the development and implementation of new models of nutrition care for adults with critical illness.

On the day of study commencement (day 1), all patients treated in the ICU and admitted to the ICU after 00:00 will be screened for eligibility. Observational data will be collected days 1 and 3 of their ICU stay (whilst present in ICU) and then days 7, 14, 21 and 28 (whether they are in ICU or the ward) as well as the first full day on the ward (day after ICU discharge).

At the completion of the project, the investigators will hold the largest sample of nutrition care in critical illness in Australia (approximately 1200 Adult patients including the pilot data period) and the only international database to include the period after ICU discharge. This proposal directly links with the National Safety and Quality Health Service (NSQHS) Standard 5 (Comprehensive Care) and Standard 2 (Partnering with Consumers) and will rapidly provide data about nutrition care and hospital acquired malnutrition (a serious reportable consequence under Standard 5) to inform the accreditation process and provide a risk mitigation strategy to prevent malnutrition before it occurs. This data will be used to improve and re-design nutrition care, as well as generate new research priorities that are highly relevant to issues within clinical care, with the potential to save millions of dollars in healthcare expenditure nationally.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Admitted to ICU after 00:00 on the date of study commencement
3. Remain in ICU for ≥ 48 hours

Exclusion Criteria:

1. Patients who have been deemed ready to be discharged by the treating team within 48 hours of ICU admission but have not been able to be discharged within 48 hours of ICU admission for logistical reasons (e.g., due to bed unavailability, inability to return home)
2. Patients who have been admitted for palliative care or organ donation or made palliative within 48 hours of ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In a 7 day study period, all adult patients present in the ICU who meet all of the inclusion criteria and no exclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Nutritional outcomes | Up to day 28 of hospitalization
  Protein and energy prescription and provision
Nutritional outcomes | Up to day 28 of hospitalization
  Use of Enteral Nutrition (EN)
Nutritional outcomes | Up to day 28 of hospitalization
  Parenteral Nutrition (PN)
Nutritional outcomes | Up to day 28 of hospitalization
  Oral intake and oral nutrition supplements
Nutrition service delivery in the ICU and ward setting | Up to day 28 of hospitalization
  Levels of staffing available and service provision for nutrition care in the ICU and on the ward
Descriptions of nutrition prescription, delivery and service variability across ANZ | Up to day 28 of hospitalization
  Comparison of nutrition care between participating hospitals
Patient-centred outcomes | Up to day 28 of hospitalization
  Duration of hospital stay
Patient-centred outcomes | Up to day 28 of hospitalization
  Mortality
Patient-centred outcomes | Up to day 28 of hospitalization
  Discharge destination

CONTACTS AND LOCATIONS:
Locations (1):
- Monash University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No